CLINICAL TRIAL: NCT06920069
Title: Phase IV Study of Evaluating Immunogenicity and Safety of Concomitant Administration of Sabin-strain-based Inactivated Poliovirus Vaccine (Vero Cells) and Adsorbed Acellular Pertussis, Diphtheria and Tetanus Combined Vaccine or Measles, Mumps and Rubella Combined Live-attenuated Vaccine
Brief Title: Study of Concomitant Administration of the sIPV and DTaP or MMR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sIPV-401
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Polio; Diphteria, Tetanus and Pertussis; MMR Vaccine
MeSH Terms: conditions — Poliomyelitis; Tetanus; Whooping Cough | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- sIPV + DTaP (concomitant vaccination cohort) (Experimental): sIPV at 2,3,4 and 18 months of age, DTaP at 2,4,6 and 18 months of age
  Interventions: Biological: sIPV; Biological: DTaP
- sIPV/bOPV + DTaP (concomitant vaccination cohort) (Experimental): sIPV at 2,3 months of age and bOPV at 4 months and 4 years of age DTaP at 2, 4, 6 and 18 months of age
  Interventions: Biological: sIPV; Biological: DTaP; Biological: bOPV 1,3
- sIPV + DTaP + MMR (systematic interval-based vaccination cohort) (Experimental): sIPV at 2,3,4 and 18 months of age DTaP at 2,4,6 and 18 months of age, 7 days after the administration of sIPV MMR at 18 months of age, randomly assigned in the concomitant administration with sIPV or 1 month after the administration of DTaP
  Interventions: Biological: sIPV; Biological: DTaP; Biological: MMR Vaccine
- sIPV/bOPV + DTaP (Systematic interval-based vaccination cohort) (Experimental): sIPV at 2,3 months of age, bOPV at 4 months and 4 years of age DTaP at 2,4,6 and 18 months of age, 7 days after the administration of sIPV
  Interventions: Biological: sIPV; Biological: DTaP; Biological: bOPV 1,3

INTERVENTIONS:
Biological: sIPV — Sabin-strain-based inactivated vaccine (Vero cells), 0.5mL for each dose
Biological: DTaP — Adsorbed acellular pertussis, diphtheria and tetanus combined vaccine, 0.5mL for each dose
Biological: bOPV 1,3 — Poliomyelitis Vaccine Type I Type Ⅲ in Dragee Candy (Human Diploid Cell), Live, 1g for each dose
  Arms: sIPV/bOPV + DTaP (Systematic interval-based vaccination cohort); sIPV/bOPV + DTaP (concomitant vaccination cohort)
Biological: MMR Vaccine — Measles, Mumps and Rubella Combined Live-attenuated Vaccine, 0.5mL for each dose
  Arms: sIPV + DTaP + MMR (systematic interval-based vaccination cohort)

SUMMARY:
This study is a randomized, open-labeled phase IV clinical trial to evaluate the immunogenicity and safety of concomitant administration of sIPV and DTaP or MMR in infants aged 2 months. Primary immunogenicity endpoints in all groups include the seroconversion rate of type I, II, and III anti-poliovirus neutralizing antibodies, anti-DT, anti-TT, anti-PT, anti-FHA, and anti-PRN antibodies 30 days after basic immunization. Secondary immunogenicity endpoints include the seropositive rates, seroconversion rates, geometric mean titer/concentration (GMT/GMC), geometric mean fold increase (GMFI) of type I, II, and III anti-poliovirus neutralizing antibodies, anti-DT, anti-TT, anti-PT, anti-FHA, and anti-PRN antibodies, and anti-measles, anti-mumps, and anti-rubella antibodies 30 days after full immunization. The secondary safety endpoints are the incidence of adverse events (AEs) within 30 minutes after each injection, the incidence of solicited local and systematic AEs in the period of solicitation after each injection, the incidence of unsolicited AEs in 30 days after each injection, the incidence of AEs in 30 days after each injection, and the incidence of serious adverse events in 6 months after administrations.

DETAILED DESCRIPTION:
This is a randomized, open-labeled, parallel phase IV clinical trial to evaluate the immunogenicity and safety of concomitant administration of sIPV and DTaP or MMR. 2640 participants aged 2 months will be randomly assigned to 4 cohorts in a ratio of 1:1:1:1. [Cohort A] 660 infants will take administration of sIPV at 2, 3, 4, 18 months of age and DTaP at 2, 4, 6, and 18 months of age. sIPV and DTaP at 2, 4, and 18 months of age will be taken concomitantly. [Cohort B] 660 infants will take administration of sIPV at 2, 3 months of age, bOPV at 4 months and 4 years of age, and DTaP at 2, 4, 6, 18 months of age. sIPV/bOPV at 2, 4 months of age will be taken concomitantly. [Cohort C] 660 infants will take administration of sIPV at 2, 3, 4, 18 months of age, DTaP at 2, 4, 6, and 18 months of age, and MMR at 18 months of age. DTaP will be taken 7 days after sIPV at 2, 4, 18 months of age. Half participants will take concomitant administration of sIPV and MMR at 18 months of age, and the rest will take them separately (MMR at 19 months of age). [Cohort D] 660 infants will take administration of sIPV at 2, 3 months of age, bOPV at 4 months and 4 years of age, and DTaP at 2, 4, 6, 18 months of age. DTaP will be taken 7 days after sIPV/bOPV at 2, 4 months of age.

For immunogenicity assessment, blood samples on Day 0 and Day 30 after basic immunization of each kind of investigational vaccine would be collected to evaluate the type I, II, and III anti-poliovirus neutralizing antibodies, anti-DT, anti-TT, anti-PT, anti-FHA, and anti-PRN antibodies, and anti-measles, anti-mumps, and anti-rubella antibodies for different groups.

For safety assessment, adverse events after each dose would be recorded through the diary and contact cards by participants' guardians to collect solicited or unsolicited AEs in periods of solicitation and nonsolicitation, respectively. From 31 days after the final dose to 6 months later, serious adverse events will be evaluated by the investigator via phone call or active reports by participants' guardians.

ELIGIBILITY:
Inclusion Criteria:

* Age Requirement: Infants aged 2 months at the time of enrollment
* Provision of Legal Identification: Volunteers and their legal guardians or appointed representatives must provide valid legal identification documents.
* Informed Consent: Legal guardians or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, and sign the informed consent form.
* Adherence: Legal guardians or appointed representatives of volunteers must be able to comply with the requirements in the study as well as complete relevant visits on time.
* Birth Condition: Full-term at birth (gestational age ≥ 37 weeks and < 42 weeks) and birth weight ≥ 2500g

Exclusion Criteria:

* Vaccination History: received vaccines containing diphtheria-tetanus-pertussis antigens, polio antigens, Hib conjugate vaccine, or 13-valent pneumococcal conjugate vaccine before enrollment.
* Those who had received blood transfusions or used blood products (except hepatitis B immunoglobulin) before enrollment.
* Recent Vaccination: Volunteers received any inactivated vaccines or subunit vaccines within 7 days (including the 7th day) prior to vaccination with the investigational vaccine, or any other live attenuated vaccines within 14 days (including the 14th day) prior to vaccination.
* Acute Illness: Volunteers have experienced acute illnesses (e.g., fever) within 3 days before enrollment, or have used antipyretic analgesics or antihistamines within 3 days.
* Allergic History: Volunteers who are allergic to any component of sIPV, bOPV, DTaP, or MMR, or who are allergic to kanamycin sulfate, kanamycin, or gentamicin sulfate, or those with an allergic constitution.
* Birth Condition: Severe neonatal diseases caused by abnormal delivery and other reasons, such as birth trauma, neonatal asphyxia, respiratory distress syndrome, neonatal intracranial hemorrhage, etc., or patients with clinically confirmed severe hyperbilirubinemia.
* Neurological and Mental Health: Volunteers with encephalopathy, convulsions, epilepsy, or other progressive neurological disorders, or those whose families have a history of genetic predisposition to convulsions or epilepsy, or a history of genetic predisposition to mental illness.
* History of Related Illness: Volunteers who have a history of poliomyelitis, pertussis, diphtheria, tetanus, measles, rubella, or mumps.
* Immune Therapy: Volunteers with immunodeficiency, weakened immune function, or those who have received immunosuppressive therapy (such as long-term systemic glucocorticoid treatment, but excluding local medications like inhalants or nasal sprays).
* Other Diseases: Volunteers with severe diseases, encompassing those in the cardiovascular system, blood and lymphatic systems, immune system, kidneys, liver, gastrointestinal tract, respiratory system, metabolism, and bones, etc.
* Participation in Other Clinical Studies: Volunteers are currently or have plans to participate in other clinical studies before enrollment.
* Investigator's Discretion: The final exclusion criterion is the investigator's discretion to determine whether a volunteer is suitable for participation in the study.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2640 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2030-07-15 (Estimated); Study Completion 2031-06-15 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-seroconversion rate of type I anti-poliovirus neutrilizing antibody | Between baseline and day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline
Immunogenicity index-seroconversion rate of type II anti-poliovirus neutrilizing antibody | Between baseline and day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline
Immunogenicity index-seroconversion rate of type III anti-poliovirus neutrilizing antibody | Between baseline and day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline
Immunogenicity index-seroconversion rate of anti-DT antibody | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<0.1 IU/ml) to seropositive (Antibody Concentration≥0.1 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rate of anti-TT antibody | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<0.1 IU/ml) to seropositive (Antibody Concentration≥0.1 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rate of anti-PT antibody | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<20 IU/ml) to seropositive (Antibody Concentration≥20 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rate of anti-FHA antibody | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<20 IU/ml) to seropositive (Antibody Concentration≥20 IU/ml), or a ≥4-fold increase from baseline.

SECONDARY OUTCOMES:
Immunogenicity index-seropositive rate of type I anti-poliovirus neutrilizing antibody | Day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seropositive will be defined as the antibody tie ≥1:8
Immunogenicity index-seropositive rate of type I anti-poliovirus neutrilizing antibody | Day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seropositive will be defined as the antibody tie ≥1:8
Immunogenicity index-seropositive rate of type II anti-poliovirus neutrilizing antibody | Day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seropositive will be defined as the antibody tie ≥1:8
Immunogenicity index-seropositive rate of type II anti-poliovirus neutrilizing antibody | Day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seropositive will be defined as the antibody tie ≥1:8
Immunogenicity index-seropositive rate of type III anti-poliovirus neutrilizing antibody | Day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seropositive will be defined as the antibody tie ≥1:8
Immunogenicity index-seropositive rate of type III anti-poliovirus neutrilizing antibody | Day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seropositive will be defined as the antibody tie ≥1:8
Immunogenicity index-geometric mean titer (GMT) of type I anti-poliovirus neutrilizing antibody | Day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean titer (GMT) of type I anti-poliovirus neutrilizing antibody | Day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean titer (GMT) of type II anti-poliovirus neutrilizing antibody | Day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean titer (GMT) of type II anti-poliovirus neutrilizing antibody | Day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean titer (GMT) of type III anti-poliovirus neutrilizing antibody | Day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean titer (GMT) of type III anti-poliovirus neutrilizing antibody | Day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type I anti-poliovirus neutrilizing antibody | Between baseline and day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type I anti-poliovirus neutrilizing antibody | Between baseline and day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type II anti-poliovirus neutrilizing antibody | Between baseline and day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type II anti-poliovirus neutrilizing antibody | Between baseline and day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type III anti-poliovirus neutrilizing antibody | Between baseline and day 30 after basic vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type III anti-poliovirus neutrilizing antibody | Between baseline and day 30 after full vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-seropositive rate of anti-DT antibody | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥0.1 IU/ml.
Immunogenicity index-seropositive rate of anti-DT antibody | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥0.1 IU/ml.
Immunogenicity index-seropositive rate of anti-TT antibody | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥0.1 IU/ml.
Immunogenicity index-seropositive rate of anti-TT antibody | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥0.1 IU/ml.
Immunogenicity index-seropositive rate of anti-PT antibody | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥20 IU/ml.
Immunogenicity index-seropositive rate of anti-PT antibody | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥20 IU/ml.
Immunogenicity index-seropositive rate of anti-FHA antibody | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥20 IU/ml.
Immunogenicity index-seropositive rate of anti-FHA antibody | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the antibody concentration≥20 IU/ml.
Immunogenicity index-geometric mean concentration (GMC) of antibody against DT | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against DT | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against TT | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against TT | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against PT | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against PT | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against FHA | Day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against FHA | Day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against DT | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against DT | Between baseline and day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against TT | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against TT | Between baseline and day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against PT | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against PT | Between baseline and day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against FHA | Between baseline and day 30 after basic vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against FHA | Between baseline and day 30 after full vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-seroconversion rate of anti-measles virus antibody | Between baseline and day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<200mIU/ml) to seropositive (≥200mIU/ml), or a ≥4-fold increase from baseline
Immunogenicity index-seroconversion rate of anti-rubella virus antibody | Between baseline and day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<20IU/ml) to seropositive (≥20IU/ml), or a ≥4-fold increase from baseline
Immunogenicity index-seroconversion rate of anti-mumps virus antibody | Between baseline and day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<100U/ml) to seropositive (≥100U/ml), or a ≥4-fold increase from baseline
Immunogenicity index-seropositive rate of anti-measles virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as antibody concentration ≥200mIU/ml
Immunogenicity index-seropositive rate of anti-rubella virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as antibody concentration ≥20IU/ml
Immunogenicity index-seropositive rate of anti-mumps virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as antibody concentration ≥100U/ml
Immunogenicity index-geometric mean concentration (GMC) of anti-measles virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean concentration (GMC) of anti-rubella virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean concentration (GMC) of anti-mumps virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean fold increase (GMFI) of anti-measles virus antibody | Between baseline and day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean fold increase (GMFI) of anti-rubella virus antibody | Between baseline and day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean fold increase (GMFI) of anti-mumps virus antibody | Between baseline and day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Safety index-incidence of adverse events | 0-30 minutes after vaccination
  Incidence of adverse events after vaccination
Safety index-incidence of solicitied adverse events | Day 0-7 or Day 0-14 after vaccination
  Incidence of solicited local and systematic adverse events after vaccination
Safety index-incidence of unsolicitied adverse events | Day 0-30 after vaccination
  Incidence of unsolicited adverse events after vaccination
Safety index-incidence of serious adverse events | From the beginning of the vaccination up to 6 months after vaccination completed
  Incidence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, Principal Investigator — Yunnan Provical Center for Disease Control and Prevention
Locations (9):
- China (9):
  - Lufeng Center for Disease Control and Prevenion, Chuxiong, Yunnan
  - Yuanmou Center for Disease Control and Prevention, Chuxiong, Yunnan
  - Wuding Center for Disease Control and Prevention, Chuxiong, Yunnan
  - Yaoan Center for Disease Control and Prevention, Chuxiong, Yunnan
  - Lancang Center for Disease Control and Prevention, Puer, Yunnan
  - Yanshan Center for Disease Control and Prevention, Wenshan, Yunnan
  - Qiubei Center for Disease Control and Prevention, Wenshan, Yunnan
  - Guangnan Center for Disease Control and Prevention, Wenshan, Yunnan
  - Mile Center for Disease Control and Prevention, Yisa, Yunnan

IPD SHARING:
Plan to Share IPD: No